CLINICAL TRIAL: NCT03801252
Title: Antibiotic Prophylaxis to Prevent Obesity-Related Induction Complications in Nulliparae at Term (APPOINT): A Pilot Randomized Controlled Trial
Brief Title: Antibiotic Prophylaxis to Prevent Obesity-Related Induction Complications in Nulliparae at Term
Acronym: APPOINT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9939
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Induction of Labor Affected Fetus / Newborn
MeSH Terms: conditions — Obesity | interventions — Cefazolin; Sodium Chloride; Azithromycin

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: One arm includes double placebo drugs that will be blinded from the investigator and participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cefazolin + Azithromycin (Experimental): Women will be randomized 1:1 to receive cefazolin 2 grams intravenously at the start of the labor induction and every 8 hours thereafter for a maximum of three doses and azithromycin 500 mg intravenously once at the start of the labor induction
  Interventions: Drug: Cefazolin; Drug: Azithromycin
- Placebo + Placebo (Placebo Comparator): Women will be randomized 1:1 to receive placebo intravenously at the start of the labor induction and every 8 hours thereafter for a maximum of three doses and placebo intravenously once at the start of the labor induction
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cefazolin — intravenous drugs used as prophylactic antibiotics
  Arms: Cefazolin + Azithromycin
Drug: Placebo — Intravenous saline
  Other Names: Saline
  Arms: Placebo + Placebo
Drug: Azithromycin — prophylactic antibiotic
  Arms: Cefazolin + Azithromycin

SUMMARY:
Obesity increases the risk of pregnancy complications, including among others puerperal infections and cesarean delivery, and risk rises with increasing body mass index (BMI). Class III obesity is an indication for delivery by 39 weeks, and these patients have a high rate of labor induction. In nulliparous women from the general population (obese and non-obese), labor induction at 39 weeks (compared to expectant management) is associated with less morbidity and a lower cesarean rate. Antibiotic prophylaxis, standard before cesarean delivery, is associated with less post-cesarean infection if azithromycin is added to the standard cefazolin. In this placebo-controlled pilot trial, investigators will estimate the parameters necessary to calculate the sample size for a planned multicenter clinical trial of prophylactic antibiotics administered at the start of labor inductions of morbidly obese nulliparous women at term.

DETAILED DESCRIPTION:
Investigators will enroll consenting women delivering at The Children's Hospital at OU Medical Center who meet enrollment criteria. Flyers will be distributed to providers to give to women who may be eligible for the study at prenatal visits, so that they may review the information prior to presenting for their induction of labor. Labor induction may be a scheduled procedure. However, many inductions occur in an unscheduled fashion due to medical or obstetric indications. Therefore, it is difficult to predict which women will ultimately require labor induction and at what gestational age they will require it, so it is not feasible to approach and consent all women during a clinic visit prior to labor induction. Distribution of flyers will allow patients to have information about the study prior to presenting for labor induction. Furthermore, unlike women in spontaneous labor, women being consented just prior to a labor induction are not vulnerable in the same way as one might consider a patient in labor, since they will not have the distraction and discomfort of uterine contractions that are presenting in laboring patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30
* No prior deliveries at or beyond 20 weeks gestation
* Undergoing induction of labor
* Gestational age 37 weeks or more
* Age 15-45

Exclusion Criteria:

* Fetal death prior to labor induction
* Known fetal anomaly
* Multiple gestation
* Ruptured membranes for more than 12 hours
* Chorioamnionitis or other infection requiring antibiotics at the start of the labor induction
* Previous myometrial surgery
* Allergy to either drug used in the protocol (cefazolin or azithromycin)

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women of child-bearing age
Enrollment: 186 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Pierce, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Pierce SL, Peck JD, Zornes C, Standerfer E, Edwards RK. Antibiotic Prophylaxis to Prevent Obesity-Related Induction Complications in Nulliparae at Term: a pilot randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Sep;4(5):100681. doi: 10.1016/j.ajogmf.2022.100681. Epub 2022 Jun 18. PMID 35728781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Researchers enrolled women delivering at The Children's Hospital at OU Medical Center who met enrollment criteria and consented to study participation. Patients were given information about the study during a third trimester prenatal care visit. However, they were enrolled in the hospital before their labor induction is started.
Period: Overall Study
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Started | 93 | 93
Completed | 92 | 91
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cefazolin + Azithromycin: Women were randomized 1:1 to receive cefazolin 2 grams intravenously at the start of the labor induction and every 8 hours thereafter for a maximum of three doses and azithromycin 500 mg intravenously once at the start of the labor induction
  Cefazolin: intravenous drugs used as prophylactic antibiotics
  Azithromycin: prophylactic antibiotic
- Placebo + Placebo: Women were randomized 1:1 to receive placebo intravenously at the start of the labor induction and every 8 hours thereafter for a maximum of three doses and placebo intravenously once at the start of the labor induction
  Placebo: Intravenous saline
- Total: Total of all reporting groups
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo | Total
Number analyzed (Participants) | 93 | 93 | 186
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (y) | 26.9 (5.6) | 25.3 (5.2) | 26.1 (5.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female participants | 93 | 93 | 186
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: White | 57 | 46 | 103
  Race and ethnicity: Black | 7 | 9 | 16
  Race and ethnicity: Hispanic | 16 | 18 | 34
  Race and ethnicity: Asian | 4 | 2 | 6
  Race and ethnicity: Native American | 7 | 11 | 18
  Race and ethnicity: Other | 2 | 5 | 7
  Race and ethnicity: Not reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 93 | 93 | 186
BMI ≥30 [Count of Participants; unit: Participants]
  Class I (BMI, 30-34 kg/m^2) | 19 | 19 | 38
  Class II (BMI, 35-39 kg/m^2) | 23 | 24 | 47
  Class III (BMI, ≥40 kg/m^2) | 51 | 50 | 101
Gestational age 37 weeks or more [Mean (Standard Deviation); unit: days] | 271.4 (8.4) | 271.7 (6.2) | 271.6 (7.3)
Chronic hypertension [Count of Participants; unit: Participants] | 9 | 8 | 17
Gestational hypertension [Count of Participants; unit: Participants] | 32 | 18 | 50
Preeclampsia [Count of Participants; unit: Participants] | 19 | 22 | 41
Diabetes mellitus [Count of Participants; unit: Participants]
  Gestational | 10 | 11 | 21
  Pregestational | 8 | 5 | 13
Fetal growth restriction [Count of Participants; unit: Participants] | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cesarean Delivery
Description: Rate at which women give birth via cesarean section
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 93 | 93
Participants | 27 | 37

2. Primary Outcome: Number of Participants With Puerperal Infections
Description: Chorioamnionitis, endometritis and/or cesarean wound infection
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 93 | 93
Participants | 8 | 9

3. Secondary Outcome: Number of Participants With Postpartum Hemorrhage
Description: Experience of postpartum hemorrhage
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 93 | 93
Participants | 16 | 16

4. Secondary Outcome: Number of Participants Who Underwent A Blood Transfusion
Description: Need of a blood transfusion
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 93 | 93
Participants | 4 | 4

5. Secondary Outcome: Number of Participants With ICU Admission
Description: Intensive care unit admission
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 93 | 93
Participants | 1 | 0

6. Secondary Outcome: Number of Participants With Maternal Hospital Readmission
Description: Maternal hospital readmission within 30 days after delivery
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 93 | 93
Participants | 1 | 2

7. Secondary Outcome: Primary Indications for Cesarean Delivery
Description: Nonreassuring fetal status, failed induction, active-phase arrest, second-stage arrest, or other
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 27 | 37
Participants
  Nonreassuring fetal status | 12 | 14
  Failed induction | 11 | 11
  Active-phase arrest | 2 | 6
  Second-stage arrest | 1 | 4
  Other | 1 | 2

8. Secondary Outcome: Neonatal Outcomes
Description: Neonatal complications
Time Frame: 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
Number analyzed (Participants) | 93 | 93
Participants
  NICU admission | 11 | 10
  Respiratory distress syndrome | 8 | 7
  Intubation required within first 72 hours | 1 | 3
  Hyperbilirubinemia requiring phototherapy | 41 | 37
  Suspected or confirmed sepsis | 11 | 8
  Culture with organisms identified | 0 | 0
  Necrotizing enterocolitis | 0 | 0
  Periventricular leukomalacia | 0 | 0
  Intraventricular hemorrhage grade III or higher | 0 | 0
  Neonatal death | 0 | 0
  Neonatal complications composite | 50 | 42

ADVERSE EVENTS:
Time Frame: 30 days after delivery
Arm/Group | Cefazolin + Azithromycin | Placebo + Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/93
Other Adverse Events (participants affected / at risk) | 4/93 | 0/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cefazolin + Azithromycin (N=93) | Placebo + Placebo (N=93)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
NICU admission (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Postpartum preeclampsia/readmission (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT03801252/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT03801252/ICF_001.pdf